CLINICAL TRIAL: NCT04286113
Title: PREDHICT: Precision Recruitment and Engagement of Diabetics and Hypertensives in Clinical Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01791-substudy
Record Dates: First submitted 2020-01-09; First posted 2020-02-26 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participants will receive non-personalized information (one-size-fits-all) diet, sleep and physical activity recommendations via messaging delivered by app.
  Interventions: Behavioral: control group
- Intervention Group (Experimental): Participants will receive personalized messages about achieving healthy diet, physical activity and sleep as well as summary of their performance for the week and month. They will also receive personalized content about research volunteerism and altruistic activities.
  Interventions: Behavioral: Lifestyle management

INTERVENTIONS:
Behavioral: control group — will receive standard medical care where research assistant will give pamphlets, with one size fits all recommendations for diet/nutrition, physical activity and sleep, to 10 subjects with comorbid HTN and T2D.
  Arms: Control group
Behavioral: Lifestyle management — Will use passive ubiquitous sensing through FitBit to 1)learn behavioral profiles of subjects who have pre-HTN/HTN and/or pre-diabetes /Diabetes 2) provide personalized recommendations through mobile based messaging app that will increase the likelihood of engaging in health diet/nutrition, physical activity and sleep practices
  Arms: Intervention Group

SUMMARY:
For the sub-study, this digital navigation tool will both inform/educate, engage, support, and navigate participants and providers through the process of clinical trial participation via personalization (data profiling, adaptive and customized messaging, and tailored digital navigation) in a sample of 100 participants with diabetes and hypertension.

DETAILED DESCRIPTION:
To identify provider- and system-level facilitators (solutions) of clinical trial participation that can be in corporated in the digital navigation tool. We will pay special emphasis on the behavior research volunteerism and altruism and individuals who are at risk for cardio metabolic conditions. To develop solutions that will address patient-, provider and system-level barriers preventing clinical trial participation Objective 2: To test the adherence, feasibility, and efficacy of a research volunteerism and altruism component of a health and wellness web app. that provides personalized newsfeeds and curriculum about research and health-related volunteer and altruistic activities versus traditional patient navigation procedures and resources in clinical trial awareness.'awareness/knowledge, attitudes, willingness to participate in clinical trial, self-efficacy, and share knowledge about clinical trial opportunities to social network. To determine which elements of the digital tool and mobil app are associated with increased awareness/knowledge, intent to participate, and contagion

ELIGIBILITY:
Inclusion Criteria:

* NYU and/or Bellevue patient
* Diagnosed with HTN and pre-diabetes/diabetes
* Must be English speakers
* Ownership of a smart phone and are willing to use it to download app built in TrialX which will be free for participants
* Must be ambulatory

Exclusion Criteria:

* are unable or unwilling to provide informed consent;
* are unable to participate meaningfully in an intervention that involves self-- monitoring using software available in English (e.g., due to uncorrected sight impairment, illiterate, non-English-speaking, dementia);
* are institutionalized (e.g., in a nursing home or personal care facility, or those who - are incarcerated and have limited control over self-management)
* have a history of heart disease, kidney disease, or retinopathy (to rule-out those with long-standing, undiagnosed T2D)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Change in clinical trials participation Change in User Adherence | Baseline Visit, 4 week follow up visit, 6 month follow up visit
  Will show that one-size-fits-all versus personalization leads to greater adherence. Adherence will be based on whether the subject met the daily and weekly behavior recommendations.
Change in glucose level Change in blood pressure | Baseline Visit, 4 week follow up visit, 6 month follow up visit
  The amount of sugar levels will be determined the Harris-Benedict Calculator, which consists of height, weight, weight age and activity levels
Change in body mass index Change in blood pressure | Baseline Visit, 4 week follow up visit, 6 month follow up visit
  Change in body mass index will be determined by the self reported information the vb=vodt
Change in physical activity | Baseline Visit, 4 week follow up visit, 6 month follow up visit
  FitBit tracking will measure increase in physical activity adherence.
Change in physical activity by self-report | Baseline Visit, 4 week follow up visit, 6 month follow up visit
  Increase in physical activity will be measured by self-report diaries collected by study staff through health and wellness app platforms.

CONTACTS AND LOCATIONS:
Overall Officials: Azizi Seixas, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: ICF
Time Frame: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided).
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.